CLINICAL TRIAL: NCT00532142
Title: A Multicenter Trial for Surgical Treatment of Central Retinal Vein Occlusion - Radial Optic Neurotomy for CVO The ROVO Study
Brief Title: The ROVO Study: Radial Optic Neurotomy for CVO
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rudolf Foundation Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EK-04-010-0204
Record Dates: First submitted 2007-09-18; First posted 2007-09-20 (Estimated); Last update posted 2009-10-30 (Estimated); Status verified 2009-10

CONDITIONS: Central Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Intravitreal Triamcinolone
Procedure: Radial Optic Neurotomy
Other: Placebo - Sham Intravitreal Injection

SUMMARY:
The ROVO study is a prospective, placebocontrolled and randomised study designed to evaluate the effect of radial optic neurotomy in central vein occlusion, versus triamcinolone acetonide. 240 patients with a visual acuity < 0.5 Snellen will be randomised. Patients are treated with either RON, or a single intravitreal injection of 4 mg triamcinolone acetonide, or a placebo treatment - a "sham" injection of intravitreal triamcinolone. Patients will be examined regularly over a period of one year.

Best corrected visual acuity for far and near, as well as clinical examinations, fluorescein- and indocyanine green angiograms, optical coherence tomography, and perimetry, are performed pre- and postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Onset of CVO not longer than 12 months
* On FLA 1. nonperfused - (greater than 10 disc area of nonperfusion) 2. perfused - visual acuity lower than 0.1 Snellen,or 3. perfused with no improvement of visual acuity over 4 weeks)

Exclusion Criteria:

* • Dense cataract* (grade 3 and 4) which precludes judgement of the fundus.

  * Pregnancy
  * Allergy against Fluoresceine or Indocyanine green
  * Unable to come for follow up visit
  * Presence of other severe retinopathy or
  * Presence of advanced optic atrophy or uncontrolled glaucoma.
  * Visual acuity higher than 0.5 Snellen.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2005-04; Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Proportion of eyes with an improvement of more than 15 letters (approximately > 3 lines of visual acuity gain) after one year as compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Binder, M.D., Study Chair — no affiliation
Locations (1):
- Rudolf foundation Clinic, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Aggermann T, Brunner S, Krebs I, Haas P, Womastek I, Brannath W, Binder S; ROVO Study Group. A prospective, randomised, multicenter trial for surgical treatment of central retinal vein occlusion: results of the Radial Optic Neurotomy for Central Vein Occlusion (ROVO) study group. Graefes Arch Clin Exp Ophthalmol. 2013 Apr;251(4):1065-72. doi: 10.1007/s00417-012-2134-1. Epub 2012 Sep 8. PMID 22960949